CLINICAL TRIAL: NCT05971329
Title: Pilot Study of ZetaFuse™ Bone Graft for the Treatment of Cervical Degenerative Disc Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zetagen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ZG-2022-003
Record Dates: First submitted 2023-07-18; First posted 2023-08-02 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-07

CONDITIONS: Radiculopathy, Cervical; Myelopathy Cervical; Neurological Abnormality; Disc Disease; Disc Degeneration
MeSH Terms: conditions — Radiculopathy; Nervous System Malformations; Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: ZetaFuse Bone Graft
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot Study of ZetaFuse Bone Graft for the Treatment of Cervical Degenerative Disc Disease (Experimental): Involves the use of a medical device. The prepared ZetaFuse Bone Graft is packed into the hollow space of a PEEK interbody before surgical implantation.
  Interventions: Device: Cervical Fusion (ZetaFuse™ Bone Graft)

INTERVENTIONS:
Device: Cervical Fusion (ZetaFuse™ Bone Graft) — Fusion of the C3-C7 cervical vertebral bodies

SUMMARY:
The goal of this pilot clinical trial is to test the safety and preliminary performance of the ZetaFuse Bone Graft in patient requiring fusion of the C3-C7 vertebral bones due to pain or loss of neurological function.

Participants will be treated with ZetaFuse during surgical intervention to reduce pain and the loss of neurological function.

DETAILED DESCRIPTION:
The indication under investigation is for use in the skeletally mature patients for fusion of one or two contiguous vertebral bodies in the cervical spine from C3-C7 following discectomy for intractable radiculopathy with or without neck pain, or myelopathy due to abnormality localized to the disc space and manifested by at least one of the following conditions confirmed by radiographic imaging:herniated nucleus pulposus, spondylosis (defined by the presence of osteophytes), and/or visible loss of disc height as compared to adjacent levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 to 75 years (inclusive) at the time of enrollment.
2. Diagnosis of radiculopathy and/or myelopathy of the cervical spine, with pain, paresthesias or paralysis in a specific nerve root distribution C3 through C7, including at least one of the following:

   * Neck and/or arm pain (at least 3 on the 0 - 10 numeric rating scale for pain.
   * Decreased muscle strength of at least one level on the clinical evaluation 0 to 5 scale.
   * Abnormal sensation including hyperesthesia or hypoesthesia. and/or
   * Abnormal reflexes.
3. Symptomatic at one or two contiguous levels from C3 to C7.
4. Radiographically determined pathology at the level to be treated correlating to primary symptoms including at least one of the following:

   * Decreased disc height on radiography, computed tomography (CT), or magnetic resonance imaging (MRI) in comparison to a normal adjacent disc.
   * Degenerative spondylosis on CT or MRI.
   * Disc herniation on CT or MRI.
5. Neck Disability Index Score ≥ 30/100.
6. Unresponsive to non-operative treatment (e.g., rest, heat, physical therapy, chiropractor, massage, pain medication) for approximately six weeks from the symptom onset; or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of continued non-operative management.
7. No previous surgical intervention at the involved levels or any subsequent, planned/staged surgical procedure at the involved or adjacent levels.
8. Appropriate for treatment using an anterior surgical approach.
9. Skeletally mature at the time of the surgery.
10. Medically cleared for surgery.
11. If a female of child-bearing potential, subject is non-pregnant, nonnursing, and agrees not to become pregnant during the study period.
12. Willing and able to comply with the study plan.
13. Signed written Patient Informed Consent Form.
14. Willing to discontinue use of non-steroidal anti-inflammatory drugs (NSAIDs) from one week before the surgery to 3 months after the surgery.

Exclusion Criteria:

1. A cervical spinal condition other than symptomatic cervical degenerative disc disease requiring surgical treatment at the involved levels.
2. Documented or diagnosed cervical instability relative to adjacent segments at either level, defined by dynamic (flexion/extension) radiographs showing sagittal plane translation >3.5 mm or sagittal plane angulation > 20°.
3. More than two cervical levels requiring surgical treatment.
4. An immobile or spontaneously fused level adjacent to the levels to be treated.
5. Severe pathology of the facet joints of the involved vertebral bodies.
6. Previous surgical intervention at either one or both of the involved levels or at adjacent levels.
7. History of trauma to the C3 to C7 levels resulting in significant bony or disco-ligamentous cervical spine injury.
8. Previously diagnosed with osteomalacia;
9. Any of the following that may be associated with an increased risk osteoporosis (if "Yes" to any of the below risk factors, a DEXA Scan is required to determine eligibility). If the level of bone mineral density (BMD) on DEXA scan is a T score of -2.5 or worse (i.e., -2.6, - 2.7, etc.) the subject is ineligible for the study.

   * Postmenopausal non-Black female over 60 years of age who weighs less than 140 pounds.
   * Postmenopausal female who has sustained a non-traumatic hip, spine, or wrist fracture.
   * Male over the age of 60 who has sustained a non-traumatic hip or spine fracture.
   * Taking bisphosphonate medication for the treatment of osteoporosis.
   * Chronic use of high dose steroids.
10. Reported active malignancy that included a history of any invasive malignancy (except non-melanoma skin cancer) unless the subject had been treated with curative intent and there had been no clinical signs or symptoms of the malignancy for at least five years.
11. Overt or active systemic infection, or infection at the operative site.
12. Insulin dependent diabetes.
13. A tobacco user who does not agree to suspend smoking prior to surgery.
14. Chronic or acute renal failure or prior history of renal disease.
15. Mentally incompetent (If questionable, obtain psychiatric consult).
16. A prisoner.
17. An alcohol and/or drug abuser currently or recently undergoing treatment for alcohol and/or drug abuse.
18. Involved with current or pending litigation regarding a spinal condition.
19. Received drugs that may interfere with bone metabolism within two weeks prior to the planned date of spinal surgery (e.g., steroids or methotrexate) excluding routine perioperative anti-inflammatory drugs.
20. A history of an endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's Disease, renal osteodystrophy, Ehlers- Danlos Syndrome, or osteogenesis imperfecta).
21. A condition that requires post-operative medications that interfere with the stability of the implant, such as steroids. (This does not include low dose aspirin for prophylactic anticoagulation and routine perioperative anti-inflammatory drugs).
22. Received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following implantation with the ZetaFuse™ Bone Graft device.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Subjects with Radiologic Determination of Bone Fusion of the Treated Cervical Vertebral Bones | 1 year post surgery
  Radiological Fusion of the cervical vertebral bones, assessed using planar X-radiographs or computed tomography. Fusion is defined as continuous bridging bone between the endplates of the operated cervical vertebral bones. Subjects with fusion will be assessed as having a successful outcome while subjects without fusion will have failed the procedure.

SECONDARY OUTCOMES:
Quality of Life via Short Form (SF12v2) Health Survey | 1 year post surgery
  SF12 measures quality of life, pain, and activity in a survey using 12 questions, with scores >50 showing a better outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Prince of Wales Public Hospital, Randwick, New South Wales

IPD SHARING:
Plan to Share IPD: No